CLINICAL TRIAL: NCT07216794
Title: Small Trial of Alendronate Impact on the Reservoir of HIV
Acronym: STAIR-HIV
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: A5428; 39123 (Other: DAIDS-ES ID)
Record Dates: First submitted 2025-10-10; First posted 2025-10-15 (Actual); Last update posted 2025-10-15 (Actual); Status verified 2025-10

CONDITIONS: HIV
MeSH Terms: interventions — Alendronate

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Arm A: Alendronate (Experimental)
  Interventions: Drug: Alendronate
- Arm B: Placebo (Placebo Comparator)
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Alendronate — 70 mg oral capsules
  Arms: Arm A: Alendronate
Other: Placebo — Matching ALN placebo oral capsules
  Arms: Arm B: Placebo

SUMMARY:
This clinical trial is designed to test the effects of alendronate (ALN) on people living with HIV who are already receiving antiretroviral therapy (ART). Participants are randomly assigned in a 2:1 ratio to either receive alendronate or a placebo, and neither the participants nor the researchers know who is receiving the actual treatment. The goal is to see if alendronate can reduce the size and activity of the HIV-1 reservoir in these individuals.

ELIGIBILITY:
Inclusion Criteria:

1. Participants must have a confirmed HIV-1 diagnosis. This can be shown by any approved rapid HIV test or HIV enzyme/chemiluminescence test done at any time before joining the study.
2. The diagnosis must be confirmed by one of the following tests: a second different antibody test, quantitative or qualitative HIV-1 RNA PCR, HIV DNA PCR, HIV total nucleic acid test, HIV-1/2 differentiation assay, or Western blot. All tests must use whole blood, serum, or plasma (not dried blood spots) and be FDA-approved if available.
3. Participants must have been on ART for at least 1 year before joining the study, with no interruptions longer than 7 consecutive days in the past 48 weeks.
4. Participants must have been on ART for no more than 10 years before joining the study.
5. Participants should not plan to change their ART regimen during the study.
6. Participants' CD4 cell count must be at least 350 cells/mm³, measured within 30 days before joining the study, at a certified laboratory.
7. Participants' HIV-1 RNA levels must be below 50 copies/mL for the past 48 weeks and for a sample taken within 30 days before joining the study, measured at a certified laboratory.
8. Participants must have the following lab values within 30 days before joining the study, measured at a certified laboratory:

   * White blood cells (WBC) ≥ 2,500 cells/mm³
   * Absolute neutrophil count (ANC) > 1,000 cells/mm³
   * Hemoglobin > 12 g/dL for males and > 11.5 g/dL for females
   * Platelet count ≥ 125,000 cells/mm³
   * Liver enzymes (AST, ALT, alkaline phosphatase) < 1.5 times the upper limit of normal (ULN)
   * Total bilirubin < 1.5 times ULN
   * Vitamin D level > 15 ng/mL
   * Estimated glomerular filtration rate (eGFR) ≥ 35 mL/min/1.73 m²
   * Negative hepatitis B surface antigen (HBsAg)
   * Negative hepatitis C antibody or RNA test
   * Calcium level between 8.4 mg/dL and 10.6 mg/dL
   * Phosphate level ≥ 3.4 mg/dL
9. If participants are women who could become pregnant, they must have a negative pregnancy test within 48 hours before joining the study. This test must be done at a certified clinic or laboratory.
10. If participants are women who could become pregnant and are sexually active, they must agree to use two methods of contraception from 10 days before starting the study until the end of the study. One method must be highly effective (e.g., implant, IUD, oral contraceptives, injectable contraceptives, vaginal ring, contraceptive patch, or sterilization of male partner). The second method must be a barrier method (e.g., condoms, diaphragm, cervical cap, or sponge with spermicide).
11. Participants must have a Karnofsky performance score of at least 70 within 90 days before joining the study.
12. If participants are postmenopausal women or men aged 50 or older, they must have a DEXA scan within 2 years before joining the study to check for osteoporosis. If participants have severe bone thinning (osteopenia), they may need another DEXA scan before joining the study.
13. Participants must be able to swallow pills without difficulty.

Exclusion Criteria:

1. Participants who started antiretroviral therapy (ART) during the early stages of HIV infection.
2. Male participants with low testosterone levels (below 250 ng/dL) within 90 days before joining the study, or those with levels between 250-400 ng/dL who plan to start testosterone replacement within 90 days before joining the study.
3. Males with stable hypogonadism who have been on the same dose of testosterone treatment for at least 24 weeks can join if they don't plan to change their regimen during the study.
4. Participants with current or past conditions that cause esophageal inflammation, ulcers, strictures, or swallowing disorders (e.g., Barrett's esophagus, scleroderma, esophageal strictures, achalasia, or other motility disorders).
5. Participants with severe, uncontrolled reflux that might increase the risk of esophagitis, according to the site investigator.
6. Participants who had esophagitis within the past year.
7. Participants with a history of Paget's disease.
8. Participants with a history of osteoporosis.
9. Participants who had a bone fracture within the past 180 days.
10. Participants who had one or more bone fractures not caused by trauma since age 18.
11. Participants with diagnosed bleeding disorders or those currently taking anticoagulants or blood factor products.
12. Participants who cannot stand up or sit upright for at least 30 minutes.
13. Participants who used systemic glucocorticoids for more than 30 days within the past 180 days at doses higher than or equivalent to 7.5 mg prednisone/day or 30 mg hydrocortisone/day.
14. Participants with active or recent cancer requiring chemotherapy, immunotherapy, or surgery within the past 36 months or expected to need such treatments in the next year.
15. Participants with advanced liver disease (non-alcoholic fatty liver disease, steatohepatitis, or alcoholic liver disease) with known or suspected cirrhosis or fibrosis score ≥F3.
16. Participants who had invasive dental procedures within the past 6 weeks or plan to have them within the next 40 weeks (regular dental cleanings are allowed).
17. Participants with significant active periodontal or other pre-existing dental disease at the time of joining the study.
18. Participants who are currently pregnant, breastfeeding, or planning to become pregnant during the study.
19. Participants who used oral complementary or alternative medicines (herbal and homeopathic products) within the past 14 days.
20. Participants who used bisphosphonates (oral or injectable) within the past 12 months.
21. Participants with known allergies or sensitivities to ALN, the components of the tablet, or bisphosphonate compounds.
22. Participants with active drug or alcohol use or dependence that would interfere with adherence to study requirements, according to the site investigator.
23. Participants with acute or serious illness requiring systemic treatment and/or hospitalization within the past 90 days.
24. Participants who received any investigational vaccine within the past 180 days or any vaccine within the past 14 days.
25. Participants who received anti-HIV broadly neutralizing antibody therapy within the past 78 weeks.
26. Participants who received a latency-reversing agent within the past 12 months, unless reviewed and approved by the A5428 Clinical Management Committee (CMC).

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2026-01-17 (Estimated); Primary Completion 2027-03-26 (Estimated); Study Completion 2027-05-21 (Estimated)

PRIMARY OUTCOMES:
Change in intact HIV-1 deoxyribonucleic acid (DNA) copies by the Intact Proviral DNA Assay (IPDA) in peripheral blood | Baseline to week 24

SECONDARY OUTCOMES:
Amount of ALN excreted after initial dose of ALN | Over 24 hours
Peripheral blood CD4+ cell-associated (CA) HIV-1 RNA levels (unspliced and multiply spliced species by quantitative polymerase chain reaction [qPCR]) | At Baseline and Weeks 12, 24 and 32
Number of plasma HIV-1 RNA copies [by single copy assay (SCA)] | At Baseline and Weeks 12, 24 and 32
HIV RNA in the GI tract (RNA scope and spatial immunophenotyping in sigmoidoscopy samples) | Pre-intervention and Weeks 22-24
Number of intact HIV-1 DNA copies by the IPDA in peripheral blood | Weeks 2, 12, and 32
HIV DNA in the GI CD4+ and Vdelta1 (Vd1) T cells (DNA scope in sigmoidoscopy samples) | Pre-intervention and Weeks 22-24
Peripheral blood CD4+ cell-associated (CA) HIV-1 RNA levels (unspliced and multiply spliced species by qPCR) | At Baseline and Weeks 1 and 2
Number of plasma HIV-1 RNA copies (by SCA) | At Baseline and Weeks 1 and 2
Frequency of αβ CD8+ cells by flow cytometry | Pre-intervention and Weeks 1, 12, 24, and 32
Phenotype of αβ CD8+ cells by flow cytometry | Pre-intervention and Weeks 1, 12, 24, and 32
Frequency of γδ cells by flow cytometry | Pre-intervention and Weeks 1, 12, 24, and 32
Phenotype of γδ cells by flow cytometry | Pre-intervention and Weeks 1, 12, 24, and 32
Frequency of NK cells by flow cytometry | Pre-intervention and Weeks 1, 12, 24, and 32
Phenotype of NK cells by flow cytometry | Pre-intervention and Weeks 1, 12, 24, and 32
HIV-specific responses (IFN- γ and GzmB) by Fluorospot | Pre-intervention and Weeks 1, 12, 24, and 32
Presence of plasma markers of inflammation/activation | Pre-intervention and Weeks 1, 12, 24, and 32

CONTACTS AND LOCATIONS:
Locations (5):
- United States (5):
  - University of California, San Francisco HIV/AIDS (Site ID: 801), San Francisco, California
  - University of Colorado Hospital (Site ID: 6101), Aurora, Colorado
  - Chapel Hill (Site ID: 3201), Chapel Hill, North Carolina
  - Ohio State University (Site ID: 2301), Columbus, Ohio
  - University of Pittsburgh (Site ID: 1001), Pittsburgh, Pennsylvania

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data that underlie results in the publication, after deidentification.
Supporting Information: Study Protocol, SAP
Time Frame: Beginning 3 months following publication and available throughout period of funding of the ACTG (Advancing Clinical Therapeutics Globally for HIV/AIDS and Other Infections) by NIH.
Access Criteria: * With whom? Researchers who provide a methodologically sound proposal for use of the data that is approved by the ACTG (Advancing Clinical Therapeutics Globally for HIV/AIDS and Other Infections).
  * For what types of analyses? To achieve aims in the proposal approved by the ACTG.
  * By what mechanism will data be made available? Researchers may submit a request for access to data using the ACTG "Data Request" form at: https://actgnetwork.org/submit-a-proposal/. Researchers of approved proposals will need to sign an ACTG Data Use Agreement before receiving the data.